CLINICAL TRIAL: NCT07190768
Title: The Comparison of the Effectiveness of Kinesiologic Taping and Dry Needling in the Treatment of Subacromial Pain Syndrome: a Randomize Trial
Brief Title: Effectiveness of Kinesiologic Taping and Dry Needling in the Treatment of Subacromial Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Erkan KAYA, Assoc. Prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-3
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome
Keywords: Kinesiologic taping; shoulder pain; dry needling
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome | interventions — Dry Needling; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kinesio Taping + Exercise (Experimental)
  Interventions: Other: Kinesio Taping; Behavioral: Exercise Program
- Dry Needling + Exercise (Experimental)
  Interventions: Other: Dry Needling; Behavioral: Exercise Program
- Kinesio Taping + Dry Needling + Exercise (Experimental)
  Interventions: Other: Kinesio Taping; Other: Dry Needling; Behavioral: Exercise Program
- Conventional Physical Therapy + Exercise (Control) (Active Comparator)
  Interventions: Behavioral: Exercise Program; Device: Conventional Physical Therapy (TENS/Ultrasound/Heat pack)

INTERVENTIONS:
Other: Kinesio Taping — Participants received Kinesio Taping (KT) applied to the affected shoulder using standard 5-cm Kinesio Tex tape. Before application, an allergy test was performed by placing a small patch of tape on the contralateral forearm for 15 minutes. The taping procedure included three regions: supraspinatus muscle, deltoid muscle, and glenohumeral joint.
  Application technique:
  Supraspinatus: Y-strip applied from insertion on the greater tubercle along the muscle to its origin with 20-25% stretch.
  Deltoid: Y-strip applied from 3 cm below insertion to the origin, with anterior and posterior tails placed along corresponding edges.
  Glenohumeral joint: I-strip applied from the coracoid process, laterally under the acromion, around the posterior deltoid edge.
  Schedule: Tape was applied at baseline (Day 0), reapplied at Day 7, and removed permanently at Day 14.
  Arms: Kinesio Taping + Dry Needling + Exercise; Kinesio Taping + Exercise
Other: Dry Needling — Participants received dry needling (DN) applied with sterile, disposable stainless-steel needles (0.30 mm × 50 mm). Target muscles included the supraspinatus, deltoideus, infraspinatus, subscapularis, and pectoralis major.
  Technique: The "fast-in, fast-out" method (Hong technique) was used. After cleaning the skin with alcohol, the needle was inserted into a palpable taut band until the first local twitch response (LTR) was elicited. The needle was moved vertically (5-10 mm) at ~1 Hz for 25-30 seconds. DN was applied for 45-60 seconds per muscle.
  Schedule: Twice per week, for 3 weeks (total of 6 sessions).
  Arms: Dry Needling + Exercise; Kinesio Taping + Dry Needling + Exercise
Behavioral: Exercise Program — All participants were instructed in a standardized home-based exercise program designed to improve shoulder mobility and stability.
  Content: Exercises included active range-of-motion movements, scapular stabilization, and strengthening of rotator cuff and periscapular muscles. Ergonomic advice and posture correction were also provided.
  Delivery: Participants were taught the program in person and instructed to perform the exercises at home.
  Schedule: Exercises were performed daily for 3 weeks, in addition to the assigned intervention for each study arm.
Device: Conventional Physical Therapy (TENS/Ultrasound/Heat pack) — Participants in this arm received conventional physical therapy modalities commonly used for the management of subacromial pain syndrome.
  Modalities: Transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound, or superficial heat pack were applied based on standard clinical practice.
  Additional care: Sessions also included passive mobilization of the shoulder into end range, scapular stabilization exercises, and ergonomic/postural advice.
  Schedule: One-hour treatment sessions, 5 days per week, for 3 consecutive weeks.
  Arms: Conventional Physical Therapy + Exercise (Control)

SUMMARY:
This study aims to compare the effectiveness of two common physiotherapy methods, Kinesiologic Taping (KT) and Dry Needling (DN), in the treatment of Subacromial Pain Syndrome (SAPS), a frequent cause of shoulder pain. The trial also investigates whether using KT and DN together provides greater benefits than using them separately. The main goal is to determine which treatment approach is more effective in reducing pain and improving shoulder function in patients with SAPS.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years

Pain in the upper, outer arm, especially during shoulder elevation

Shoulder pain lasting more than 6 weeks with or without partial rotator cuff tear

At least three of the following findings:

Painful arc during flexion or abduction

Positive Neer test

Positive Hawkins-Kennedy test

Painful resisted external rotation

Positive Jobe's test

Diagnosis confirmed by MRI evaluation when indicated

Exclusion Criteria:

Participation in a physical therapy program or receipt of injection therapy within the past 3 months

Previous shoulder surgery

Presence of joint contracture

Complete tendon rupture

Cervical radiculopathy

Systemic inflammatory disease (e.g., rheumatoid arthritis, ankylosing spondylitis)

Known allergy to tape or materials used in interventions

Bleeding disorders

Local infection or open wound in the treatment area

Cognitive dysfunction that prevents cooperation

History of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Visual Analogue Scale, VAS) | Baseline, immediately after first treatment, 1 week after first treatment, and at the end of week 3.

SECONDARY OUTCOMES:
Shoulder function (Quick-DASH questionnaire) | Baseline, 1 week after first treatment, and at the end of week 3.
Kinesiophobia (Tampa Scale of Kinesiophobia, TSK-19) | Baseline, 1 week after first treatment, and at the end of week 3.

IPD SHARING:
Plan to Share IPD: Undecided